CLINICAL TRIAL: NCT05223855
Title: 'Effect of Aquatic Physiotherapy for People With Stress; a Randomized Controlled Trial (RCT)'
Brief Title: Effect of Aquatic Physiotherapy for People With Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: vandfys (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Lone Nedergaard, Physiotherapist, vandfys
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0221
Record Dates: First submitted 2021-12-29; First posted 2022-02-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2023-09

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Intervention group receives intervention twice a week for 8 weeks. Control group receives usual care through GP for 8 weeks, and are then offered participation in de-stress class twice a week for 8 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participant is presented a numbered, opaque, sealed envelope. The outcomes assessor will be presented with data masked from group participations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group receives intervention for 8 weeks
  Interventions: Other: Physiotherapeutic hydrotherapy treatment
- control group (No Intervention): The control group receives usual care for 8 weeks and is then offered participation in a de-stress class for 8 weeks.

INTERVENTIONS:
Other: Physiotherapeutic hydrotherapy treatment — Physiotherapeutic hydrotherapy treatment The intervention consists of physiotherapeutic one-on-one treatment in a 34-36 degrees centigrade hot water, where the participants are placed supine in the water supported by the physiotherapist as well as buoyant aqua noodles. The physiotherapist supports and moves the participants in the water and adapts to the participant's reaction.
  The combination of heat, water, movement and touch affects the musculoskeletal and neuromuscular systems and thus has a depth-relaxing effect (Schoedinger, 2010).
  Arms: Intervention group

SUMMARY:
Brief summary:

Effect of aquatic physiotherapy for people with stress; a randomized controlled trial (RCT)

The purpose of the project is to investigate the effect of aquatic physiotherapy treatment in 34-36 degrees warm water.

The study is a randomized controlled trial, and participants are recruited from GPs in Lyngby-Taarbæk as well as Gentofte Kommune.

The participants are randomized using numbered, opaque and sealed envelopes.

Method:

The intervention Aquatic physiotherapy 1: 1 treatment in 34-36 degrees centigrade warm water.

The participant is placed supine in the water, supported by the physiotherapist as well as aqua noodles. The physiotherapist supports and moves the participant in the water and adapts to the participant's reaction.

Intervention Group:

The intervention group is treated twice a week. Duration of each treatment is 30 minutes. Period of treatment is 8 weeks.

Control Group:

The control group receives usual care through their GP for 8 weeks. Then they are offered participation in a de-stress class in 34-36 degrees centigrade warm water, twice a week.

Duration of each treatment is 30 minutes. Period of treatment is 8 weeks.

EFFECT MEASURES:

1. Primary effect measures:

   Change of stress level from baseline using validated questionnaire Cohen's Perceived Stress Scale (PSS).
2. Secondary effect measures:

Change of sleep disorders from baseline using validated questionnaire Pittsburgh Sleep Quality Index (PSQI).

Measurements to be taken before and after 8-weeks intervention

DETAILED DESCRIPTION:
Stress is a growing public health issue and the health professional offerings are varied and with modest evidence. Warm water has been used for centuries for the relaxing and positive effect on well-being. The evidence of this form of treatment for stress sufferers has not previously been studied.

The purpose of the project is to investigate the effect of physiotherapeutic 1:1 treatment in 34-36 degree centigrade warm water, twice a week for 30 minutes over an eight week period.

Hypothesis:

Stress sufferers will experience a reduction in stress levels.

Methodical approach:

Design: randomized controlled trial with intervention group receiving treatment in warm water and control group receiving usual care via general practitioner during the control period and then offered participation in a de-stress class.

Control group Standard treatment cf. https://www.sundhed.dk/sundhedsfaglig/laegehaandbogen/sundhedsoplysning/sundhedsoplysning/diverse/stress/

Recruitment The participants are recruited from general practitioners in Gentofte and Lyngby Tårbæk municipality, cf. inclusion and exclusion criteria.

Estimated sample sizes:

N = 26 N per group =13

Empiri:

1. Primary effect measures:

   Change of stress level from baseline using validated questionnaire Cohen's Perceived Stress Scale (PSS).
2. Secondary effect measures:

   1. Change of sleep disorders from baseline using validated questionnaire Pittsburgh Sleep Quality Index (PSQI).
   2. Change in self-perceived quality of life measured by questionnaire (EQ-5D)

   Measurements to be taken before and after 8-weeks intervention
3. Explorative measures:

a )change in self-perceived level of depression measured by questionnaire Major Depression Index (MDI), and b) change in self-perceived level of burnout measured by questionnaire Karolinska Exhaustion Disorder Scale (KEDS)

Ethical considerations:

Participation in warm water treatment is considered without side effects or risks.

Using exercise in warm water is part of general physiotherapeutic practice. The treatment is handled by experienced physiotherapists. The project complies with the Helsinki Declaration.

ELIGIBILITY:
Inclusion criteria:

* Has been reported sick by GP within the last four weeks, and is now on sick leave with stress.
* Is 18 years or older.
* Is on sick leave from work or school
* Speaks, reads and understands Danish fluently.
* Has had symptoms of stress during the last month
* Is willing to fill out questionnaires before, during and after treatment/treatment period.
* Has the possibility to participate
* Would like treatment in hot water
* Has given informed consent

Exclusion criteria:

* Previously been on sick leave with stress.
* Long-term / unresolved cases with authorities or former partners / spouses.
* Is taking sleep medication.
* Known with bipolar disorder.
* Fear of water.
* Fear of getting ears under water
* Physical state that prevents movement in water

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Level of stress | 8 weeks
  Cohens 10-item Perceived Stress Scale. A self-reported questionnaire of 10 questions that measures to which extent the respondent experiences that life is unpredictable, uncontrollable and overwhelming. Each question yields a score ranging from 0 to 4, with 4 indicating the highest level. The scores are summed to yield a total score ranging from 0 to 40 Minimum value is 0 Maximum value is 40
  The aim of the evaluation is therefore to assess whether the respondent experiences a reduction in the degree of stress.

SECONDARY OUTCOMES:
Sleep disorder | 8 weeks
  Pittsburgh Sleep Quality Index. A self-reported questionnaire that contains 19 sleep components. Each component yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  Minimum value is 0 Maximum value is 21
  The aim of the evaluation is therefore to assess whether the respondent experiences an improvement in sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bogh Juul, phD, Principal Investigator — Herlev & Gentofte Hospitalers Forskningsenhed
Locations (1):
- Lions Kollegiets varmtvandsbassin, Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The individuel participant data will not be made available to other researchers.